CLINICAL TRIAL: NCT05372146
Title: Great Saphenous Vein Sparing Segmental Radiofrequency Ablation in Varicose Veins Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 192
Record Dates: First submitted 2022-05-03; First posted 2022-05-12 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2019-11

CONDITIONS: Varicose Veins; Varicose Veins of Lower Limb
Keywords: varicose veins; chiva; hemodynamic correction
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Intervention Model Description: This was a single-center, prospective, non-randomized, non-inferiority comparative study conducted on patients with primary varicose veins
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHIVA group (Experimental): 43 participants. In the study group patients GSV was punctured 20-25 cm below SFJ. Radiofrequency catheter (ClosureFast) was inserted and positioned at SFJ distally to the superficial iliac circumflex vein. Four cycles were used for one segment below SFJ. After that catheter cooled down to 40C and was extracted. Phlebectomy was performed using Varady hooks after thermal ablation in both groups. All procedures were performed under tumescent anesthesia.
  Interventions: Procedure: GSV radiofrequency ablation with concomitant phlebectomy
- Control group (Active Comparator): 43 participants. In the controls GSV was punctured at a distal part of a refluxing segment. Catheter was positioned at SFJ and conventional radiofrequency procedure was performed with four cycles below SFJ and two cycles for every next segment. Phlebectomy was performed using Varady hooks after thermal ablation in both groups. All procedures were performed under tumescent anesthesia.
  Interventions: Procedure: GSV radiofrequency ablation with concomitant phlebectomy

INTERVENTIONS:
Procedure: GSV radiofrequency ablation with concomitant phlebectomy — Radiofrequency ablation with concomitant phlebectomy

SUMMARY:
86 patients were randomized into hot-CHIVA (n=43) and control (n=43) groups. Study group patients had undergone radiofrequency ablation (RFA) VNUS Closure - FastTM of one segment of GSV close to saphenofemoral junction. Controls had undergone whole refluxing trunk ablation. Additional phlebectomy was performed in all the patients of both groups. Primary end-point was change in quality of life (QoL) measured with CIVIQ-20 at 12 months. Secondary end-points was recurrence of varicose veins at 12 months. The investigators also measured GSV caliber at the median and distal thigh change in hot-CHIVA group.

DETAILED DESCRIPTION:
Aim - to compare GSV segmental radiofrequency ablation (hot-CHIVA) and conventional GSV ablation in varicose veins patients.

This was a single-center, prospective, non-randomized, non-inferiority comparative study conducted on patients with primary varicose veins. In a study group (hot-CHIVA) GSV segmental ablation with concomitant phlebectomy was performed. Conventional GSV radiofrequency ablation was performed in a control group. Patients were enrolled from November, 2019 to February, 2021.

All patients were examined clinically. Age, height, weight, body mass index, gender, side of disease, personal history of varicose veins were recorded. Medical history was taken. Disease description was made using advanced CEAP classification. Quality of life was measured by CIVIQ-20 and leg discomfort related to CVD symptoms on the operated leg was measured with a 10-cm visual analogue scale (VAS). Duplex ultrasound was performed in a standing position to access deep veins and GSV. We recorded reflux extention and presence of the re-entry perforators on the thigh or upper calf. Diameter of GSV near SFJ, at the middle, and lower part of the thigh was measured at inclusion in the both groups.

Sample size The sample size was calculated considering the average values for the CIVIQ-20 quality of life questionnaire on 2nd year after the endovascular treatment and CHIVA treatment obtained by reviewing the literature. Selected parameters: first-order error (α) 5%; power 80%; boundaries of "non-inferiority limit" 2; the expected difference between the study groups of 0. Taking into account the possible dropout of patients from the study, the size of the groups is increased by 5%. The estimated sample size is 86 participants.

Statistical analysis Data are presented using descriptive statistics. Normally distributed data are presented as mean with standard deviation. Not normally distributed data are presented as (Me) and interquartile range (Q1 - Q3). Two independent groups were compared with Student's t-test or Mann-Whitney test depending on data distribution. Friedman test was used to compare dependent variables. Pearson's chi-squared test or Fisher's exact test were used to compare nominal variables. A p-value of <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* C2EpAsPrGSVa, C2,3EpAsPrGSVa
* Reflux not lower than upper part of the calf,
* Age more than 18 years,
* SFJ diameter less than 15mm,
* Incompetence of terminal-femoral valve,
* GSV reflux more than 0,5 sec,
* re-entry perforator on the thigh or upper part of the calf for patients in the hot-CHIVA group

Exclusion Criteria:

* C4-C6 class of CEAP
* Pregnancy
* Deep vein reflux more than 1 sec
* SSV reflux more than 0,5 sec
* Interventions for VVs prior to the inclusion
* Those unwilling to sign an informed consent were also included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2022-02-27 (Actual)

PRIMARY OUTCOMES:
Quality of life (QoL) was measured by ChronIc Venous Insufficiency Quality of Life (CIVIQ-20) | 12 months
  There are 20 questions in the CIVIQ-20, each with 5 possible answers (1 to 5), the minimum possible score being 20 and the maximum 100. In order to calculate the GIS, the difference between the final score and the minimum possible score is to be divided by the difference between the theoretical maximum and minimum scores (100-20=80), multiplied by 100.

SECONDARY OUTCOMES:
Varicose veins recurrence | 12 months
  Visual recurrence of varicose veins
Leg discomfort related to CVD symptoms measured with 10-cm visual analogue scale (VAS) at 3 months | 2nd day, 7th day, 1 months, 3 months
  Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100.
  The following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).
In a study group remained GSV trunk diameter at mid- and lower thigh was measured at 1, 3, 6, 12 months after procedure | 1 months, 3 months, 6 months, 12 months
  Diameter of GSV measured by ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Veronika Golovina, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No